CLINICAL TRIAL: NCT02595177
Title: Multifocal Intraocular Lens vs. Monovision vs. Hybrid Monovision After Bilateral Cataract Surgery
Brief Title: Multifocal Intraocular Lens x Monovision x Hybrid Monovision After Bilateral Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Alcon Research (Industry); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Joao Crispim, Post graduated, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PresbyIOL
Record Dates: First submitted 2015-10-27; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Cataract; Presbyopia
Keywords: multifocal IOL; monovision; hybrid monovision; spectacles independence
MeSH Terms: conditions — Cataract; Presbyopia | interventions — Cataract Extraction; Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Multifocal IOL (Experimental): Cataract removal with topical anesthesia and phacoemulsification is performed. At the end, multifocal intraocular lens implantation in both eyes planning for emmetropia complete the intervention.
  Interventions: Procedure: Cataract surgery with intraocular lens implantation.
- Monovision (Experimental): Cataract removal with topical anesthesia and phacoemulsification is performed. At the end, a monofocal intraocular lens implantation planning for emmetropia in one eye (dominant) and a monofocal IOL planning for 1.50 D of myopia in the other eye (non-dominant) complete the intervention.
  Interventions: Procedure: Cataract surgery with intraocular lens implantation.
- Hybrid Monovision (Experimental): Cataract removal with topical anesthesia and phacoemulsification is performed. At the end, a monofocal intraocular lens implantation in the dominant eye and a multifocal IOL in the non-dominant eye complete the intervention.
  Interventions: Procedure: Cataract surgery with intraocular lens implantation.

INTERVENTIONS:
Procedure: Cataract surgery with intraocular lens implantation. — Phacoemulsification under topical anesthesia with intraocular lens implantation.

SUMMARY:
To compare refractive outcomes and patient's visual quality after bilateral cataract surgery when implanting multifocal intraocular lens, monofocal with monovision or hybrid monovision.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the results in randomized patients that receive bilateral multifocal IOLs, monofocal IOLs with monovision with emmetropia in one eye and 1.50 D of myopia in the other eye, or monofocal IOL in the dominant eye and multifocal IOL in the non-dominant eye, then evaluate visual and refractive outcomes, as well as independence for glasses after bilateral surgery with 1 year of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral senile cataracts.
* Implantation of IOL in the capsular bag;
* Implants from 10-30 diopter;
* Potential Visual Acuity in ≥ 0.2 logMAR (20/32, metric scale) after surgery;

Exclusion Criteria:

* Amblyopia;
* Single Eye;
* History of intraocular surgery in the previous year;
* Sequel to prior ocular trauma;
* Important Microphthalmia or aniridia;
* History of damage to the corneal endothelium (chemical burns, herpetic keratitis, corneal guttata);
* Corneal astigmatism > 1.0 D;
* IOP ≥ 21 mmHg in standard caliper;
* Ocular pathology that affects visual function (uveitis, diabetic retinopathy, age-related macular degeneration, macular dystrophy, retinal detachment, glaucoma, optic neuropathy);
* Pupil > 5 mm or < 2 mm under photopic conditions;
* Asymmetrical pupils in the eye or between the eyes;
* Binocular vision absence;
* Any situation that endangers the implant position in the capsular bag (post-traumatic zonular weakness, pseudoexfoliation, for example);
* Patient probably need to laser treatment of the retina;
* Patients whose expectations are unrealistic;
* Patients whose lifestyle involves high expectations of visual acuity (writer, driver, for example);
* Patients at risk of not meeting the clinical follow-up requirements (distance of travel difficulties, for example);

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  Binocular visual acuity in a semi-darkened room without correction to far, intermediate and near using a typical Snellen chart that is frequently used for visual acuity testing.

SECONDARY OUTCOMES:
Speed reading measure | 1 year
  Assessment is performed to measure the speed reading in each group and compare them. Then using a timer to measure how long does it take to read the page. The speed reading is measured in words per minute (WPM).
Near stereopsis measure | 1 year
  Calculate stereopsis in each group and compare them. Stereoacuity is measured using a stereogram in which separate panels are shown to each eye.
Contrast sensitivity measure | 1 year
  Comparison between groups of the contrast sensitivity. Contrast sensitivity function at five spatial frequencies is measured with the validated instrument (Functional Vision Analyzer® (Stereo Optical, Chicago, IL, USA) with best refraction.
National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25) questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joao Crispim, MD, Principal Investigator — Post graduated
Locations (1):
- Department of Ophthalmology and Visual Sciences from the Federal University of Sao Paulo (UNIFESP), São Paulo, São Paulo, Brazil